CLINICAL TRIAL: NCT05368792
Title: Prospective Trial Of Osmolar Protocol Solution on Colonoscopy Outcomes and Patient Experience
Acronym: POOPSCOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Health Centre Toronto (Other)
Collaborators: Enhanced Medical Nutrition (Industry)
Responsible Party: Principal Investigator, Ian Bookman, Gastroenterologist; Assistant Professor, St. Joseph's Health Centre Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB 21-198
Record Dates: First submitted 2021-10-29; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Colonoscopy
Keywords: Fasting; Pre-Operative Carbohydrate; Discomfort; Hydration; Bowel preparation; Bowel visibility
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The principal investigator, clinic staff and outcome assessors of colon visibility and hydration will be blinded to the treatment allocation of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex Carbohydrate (Experimental): Participants in the intervention group will be instructed to follow standard bowel preparation guidance AND consume two servings of the complex CHO (12.5% maltodextrin) drink (PREcovery®, Enhanced Medical Nutrition, Toronto, Canada) the evening prior to the procedure, and one serving 2-3 hours prior to the colonoscopy. Participants should not consume anything within 2 hours prior to the procedure's start time. One serving consists of one package (50 g maltodextrin) stirred into 400 mL of cold water.
  Standard bowel preparation guidance is as follows a split-dose 2L PEG ± bisacodyl (iso-osmolar) solution (Bi-PegLyte®, Pendopharm, Montreal, Canada) taken according to the physician's order. All participants will be instructed to follow a clear fluid diet starting the day before the procedure. Participants will also be verbally instructed to consume 2L of clear liquids the day before their colonoscopy in addition to the PREcovery.
  Interventions: Dietary Supplement: Complex Carbohydrate (PREcovery)
- Fasting (No Intervention): The Fasting arm will follow the current standard of care for colonoscopy preparations in Ontario, Canada. This includes fasting from midnight before the procedure and following a PEG bowel preparation
  All participants will follow a standard bowel preparation guidance, a split-dose 2L PEG ± bisacodyl (iso-osmolar) solution (Bi-PegLyte®, Pendopharm, Montreal, Canada) taken according to the physician's order. All participants will be instructed to follow a clear fluid diet starting the day before the procedure. Participants will also be verbally instructed to consume 2L of clear liquids the day before their colonoscopy. Participants in the fasting arm will be instructed to not have any oral intake after 00:00 of the day of their colonoscopy.

INTERVENTIONS:
Dietary Supplement: Complex Carbohydrate (PREcovery) — Each serving of the complex carbohydrate drink is a clear, colorless, 12.5% maltodextrin drink with a citrus taste, prepared by mixing 54 g of powder (50g carbohydrate) with 400mL of cold water. Participants will consume 2 servings of the complex carbohydrate drink the evening before colonoscopy (100g carbohydrate, 800mL fluid), and 1 serving 2 hours before their colonoscopy (50g carbohydrate, 400mL fluid)
  Arms: Complex Carbohydrate

SUMMARY:
Fasting is the current standard of care for colonoscopies. Recent changes to anesthesia guidelines have allowed for clear fluids to be provided up to 2 hours before procedures, including colonoscopies.

This study will compare fasting to a 12.5% carbohydrate solution 2 hours before colonoscopy on patient-reported measures of discomfort, hydration, and colon visibility.

The investigators hypothesize that the carbohydrate solution will improve patient-reported measures of discomfort, hydration, and colon visibility.

DETAILED DESCRIPTION:
Fasting and bowel preparation before colonoscopy procedures has been the clinical protocol for decades. Evidence suggests that patients undergoing this traditional standard of care before procedures may be associated with common undesirable outcomes, including anxiety, thirst, and poor patient experience. The impacts of fasting and poor satisfaction can create a cascade of challenges regarding communication between clinicians and patients.

The new standard of care utilizes an innovative clear fluid protocol, allowing patients to consume clear fluids up to 2-3 hours prior to their procedure. The consumption of a complex carbohydrate (CHO) drink may reduce dehydration, improve patient-reported outcomes, enhance patient communication and clinician workflow, ultimately resulting in improved patient experience and cancer screening/detection. Although clinical validation and implementation of a complex CHO drink have already been completed in surgical patients within clear fluid protocols, this needs to be expanded to patients undergoing colonoscopy procedures.

A prospective, single-blinded, single-centre, randomized control design will be used to compare fasting from midnight the day of the colonoscopy [the current standard of care] to a clear fluid protocol [a complex CHO drink consumed the night before and 2 hours before the colonoscopy]. The physician performing the colonoscopy will be blinded to the group allocation. The primary outcome of the present study is pre and post-procedure patient-reported measures of discomfort in adults undergoing routine colonoscopy for cancer screening. Secondary outcome measures are compliance, hydration, and bowel visibility.

Hypotheses

1. Patient-reported measures of discomfort pre and post colonoscopy will be lower in patients in the clear fluid group than the standard of care group.
2. Hydration status will be greater in the clear fluids group than the fasting group.
3. Colon visibility score (BBPS) will be higher in the clear fluids group

ELIGIBILITY:
Inclusion Criteria:

* referred for a routine colonoscopy for cancer screening
* Physician indicates a bowel preparation of split dose 2L PEG ± bisacodyl (iso-osmolar) solution

Exclusion Criteria:

* patients with colonic resection, inflammatory bowel disease; any condition that would preclude colonoscopy of the whole colon;
* patients with lower gastrointestinal bleeding, patients with ileus, gastric retention, intestinal perforation, gastrointestinal obstruction;
* patients with significant heart disease, impaired renal function, decompensated liver disease
* patients who have diabetes
* patients on opioid medications.
* Patients with a corn allergy, or allergy to any ingredient in the complex CHO drink

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Pre-procedure Patient Reported Discomfort | 30 minutes before the colonoscopy
  Domains of discomfort will be evaluated by digital VAS: anxiety, depression, hunger, inability to concentrate, malaise, nausea, pain, thirst, tiredness, unfitness, and weakness. Visual analogue scales (VAS) will be used to measure each domain. the VAS will be measured from 1-10 representing "not at all _____" and "Very ____" respectively.

SECONDARY OUTCOMES:
Hydration | Blood samples will be collected from participants immediately after the colonoscopy has ended (time point 30 minutes) and they are cleared to leave the clinic
  Plasma osmolality will be used to measure hydration status.
Compliance | 30 minutes before the colonoscopy
  Patients in the Treatment group will report the number of 50g maltodextrin packets they consumed before the procedure. Those having consumed all 3 packets provided will be reported as having 100% compliance. If the consumed none of the packets they will get a score of 0% compliance. 1 packet will result in a compliance score of 33%. 2 packets will result in a compliance score of 66%.
Bowel Visibility | During the colonoscopy (Time point 0)
  The Boston Bowel Preparation Scale (BBPS) will be used to evaluate visibility during the colonoscopy. The scale uses a 0-3 rating where 0 is the worst visibility rating ("inadequate") and 3 is the best visibility rating ("excellent"). Each of the 3 sections of the colon (left, transverse, and right) are rated using this scale and a cumulative score is determined from the sum of these three ratings.
Post-procedure Patient Reported Discomfort | up to 6 hours after the colonoscopy visit
  Domains of discomfort will be evaluated by digital VAS: anxiety, depression, hunger, inability to concentrate, malaise, nausea, pain, thirst, tiredness, unfitness, and weakness. Visual analogue scales (VAS) will be used to measure each domain. the VAS will be measured from 1-10 representing "not at all _____" and "Very ____" respectively.

IPD SHARING:
Plan to Share IPD: No